CLINICAL TRIAL: NCT05966428
Title: The Affect of Sensory Integration Therapy and Conventional Exercise Therapy on Spasticity, Balance and Motor Function With Spastic Diplegic Cerebral Palsy
Brief Title: Sensory Integration Therapy and Cerebral Palsy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Kirsehir Ahi Evran Universitesi (Other)
Responsible Party: Principal Investigator, Atahan TURHAN, Principal Investigator: Atahan Turhan, PhD, Kirsehir Ahi Evran Universitesi
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: KAEU-T.ATAHAN-001
Record Dates: First submitted 2023-07-13; First posted 2023-07-28 (Actual); Last update posted 2023-07-28 (Actual); Status verified 2023-07

CONDITIONS: Cerebral Palsy
Keywords: Sensory Integration; Physical Therapy and Rehabilitation
MeSH Terms: conditions — Cerebral Palsy

STUDY DESIGN:
Intervention Model Description: The study consisted of 2 groups as control and experiment.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control Group (Active Comparator): Conventional Exercises
  Interventions: Other: Conventional Exercises
- Intervention Group (Experimental): Conventional Exercises + Sensory Integration Therapy
  Interventions: Other: Conventional Exercises; Other: Sensory Integration Therapy

INTERVENTIONS:
Other: Conventional Exercises — This conventional exercises included stretching and strengthening, balance-coordination, mobility and range of motion exercises.
  The control group received conventional therapy 3 days a week for 8 weeks. Each therapy session a day lasted 45 minutes in control group.
Other: Sensory Integration Therapy — The Sensory Integration Therapy was applied to the intervention group in addition to the conventional exercise program. Sensory Integration Therapy included tactile, proprioceptive, and vestibular activities. The tactile sensory activities consisted of materials such as stepping stones, tactile box, brushing, fabric walking path. The vestibular sensory activities consisted of materials such as hammock swings, trampolines, rope nets, rock walls, river stones. Proprioceptive sensory activities consisted of materials such as weight bearing activities, heavy lifting, deep pressure, big ball activities, tug of war and ball pits.
  The intervention group underwent each session 45 minute conventional therapy and 15 minutes SIT. The therapy program continued 3 days a week for 8 weeks in intervention group.
  Arms: Intervention Group

SUMMARY:
This intervention study was planned to investigate the effects of Sensory Integration Therapy that added to the conventional therapy program on spasticity, balance, motor function and functional independency levels of children with spastic diplegic cerebral palsy

DETAILED DESCRIPTION:
Cerebral Palsy is a disease that can cause motor skill and posture disorders due to a non-progressive lesion in the brain that has not yet completed its development. Cerebral palsy is among the most common causes of disability in childhood. There are many conditions that can cause Cerebral Palsy. Risk groups that cause brain damage can be considered as prenatal, perinatal and postnatal risk factors.The lesion that occurs in the central nervous system in patients with Cerebral Palsy causes some problems in the musculoskeletal system, nervous system and sensory systems. In addition to these problems, depending on the level of the lesion, posture, movement disorders and balance problems occur in individuals with Cerebral Palsy. Sensory integration therapy is a neurological process of perceiving, interpreting and organizing our senses for an effective integration of the individual with the environment. When the literature is examined, the number of studies investigating the effect of sensory integration program in children with spastic diplegic type Cerebral Palsy is insufficient. The aim of this study is to investigate the effect of sensory integration therapy on spasticity, balance and motor function in children with spastic diplegic type Cerebral Palsy and to provide the data obtained at the end of the study to the literature both theoretically and practically.

The hypothesis of the study is:

* Sensory integration program reduces spasticity in children with spastic diplegic type Cerebral Palsy.
* Sensory integration program increases balance in children with spastic diplegic type Cerebral Palsy.
* Sensory integration program increases motor function in children with spastic diplegic type Cerebral Palsy.

ELIGIBILITY:
Inclusion Criteria:

* Between the ages of 4-17
* Diagnosed with spastic diplegic type Cerebral Palsy
* Having Gross Motor Function Classification System levels I and II

Exclusion Criteria:

* Children who underwent phenol and botulinum toxin-a injections in the last 6 months before the study
* Had a previous surgical operation, and had a cardiopulmonary disease that could prevent exercise
* Children with communication, hearing and vision problems

Ages: 4 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 24 (Actual)
Dates: Start 2018-01-01 (Actual); Primary Completion 2018-05-01 (Actual); Study Completion 2018-06-01 (Actual)

PRIMARY OUTCOMES:
Muscle Tone | A day before the rehabilitation
  Modified Ashworth Scale (The muscle tone evaluated on this scale is graded between 0 and 4 and is scored between 0 and 5)
Muscle Tone | 8 week
  Modified Ashworth Scale (The muscle tone evaluated on this scale is graded between 0 and 4 and is scored between 0 and 5)
Functional Balance | A day before the rehabilitation
  Pediatric Berg Balance Scale (The scale consists of 14 section. Each section is scored from 0 lowest function to 4 highest function. )
Functional Balance | 8 week
  Pediatric Berg Balance Scale (The scale consists of 14 section. Each section is scored from 0 lowest function to 4 highest function.)
Gross Motor Function | A day before the rehabilitation
  Gross Motor Function Measure (The scores are in 4 categories as "0" not starting the activity, starting independently "1", partially completing "2" and independently completing "3".)
Gross Motor Function | 8 week
  Gross Motor Function Measure (The scores are in 4 categories as "0" not starting the activity, starting independently "1", partially completing "2" and independently completing "3".)
Functional Independence | A day before the rehabilitation
  Functional Independence Measure for Children (These items are scored from 1 to 7 according to whether they received help while performing each function)
Functional Independence | 8 week
  Functional Independence Measure for Children (These items are scored from 1 to 7 according to whether they received help while performing each function)

SECONDARY OUTCOMES:
Gross Motor Function Classification | A day before the rehabilitation
  Gross Motor Function Classification System (Children with Cerebral Palsy are classified in 5 levels (1-5) according to their motor skills, functional abilities, assistive technology and wheelchair requirements)
Gross Motor Function Classification | 8 week
  Gross Motor Function Classification System (Children with Cerebral Palsy are classified in 5 levels (1-5) according to their motor skills, functional abilities, assistive technology and wheelchair requirements)

CONTACTS AND LOCATIONS:
Overall Officials: Atahan TURHAN, PhD, Principal Investigator — Kirsehir Ahi Evran University
Locations (1):
- Atahan TURHAN, Kırşehir, Merkez, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Kantor J, Hlavackova L, Du J, Dvorakova P, Svobodova Z, Karasova K, Kantorova L. The Effects of Ayres Sensory Integration and Related Sensory Based Interventions in Children with Cerebral Palsy: A Scoping Review. Children (Basel). 2022 Apr 1;9(4):483. doi: 10.3390/children9040483. PMID 35455527
- [Result] Warutkar VB, Krishna Kovela R. Review of Sensory Integration Therapy for Children With Cerebral Palsy. Cureus. 2022 Oct 26;14(10):e30714. doi: 10.7759/cureus.30714. eCollection 2022 Oct. PMID 36439588